CLINICAL TRIAL: NCT07110428
Title: Supraglottic Jet Oxygenation Ventilation During Hysteroscopic Surgery: A Randomized Controlled Trial
Brief Title: Supraglottic Jet Oxygenation Ventilation During Hysteroscopic Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-115
Record Dates: First submitted 2025-06-25; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Hysteroscopic Surgery
Keywords: SJOV; Anesthetic ventilation methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NC group (Active Comparator): Received the medication regimen: propofol at 1.5-3.0 mg/kg for sedation and fentanyl at 1.5mcg/kg for analgesia. During the maintenance phase, propofol was administered via infusion at a dose of 5 mg/kg/h . The level of sedation was maintained at 0 ≤ MOAA/S score ≤ 1. When the MOAA/S score of the subjects reached 0 after induction, nasal cannula was administered according to the group assignment. Intraoperative vital signs were closely monitored, and data on surgery duration, anesthetic dosage, blood oxygen saturation, recovery time, and possible adverse events (significant increases or decreases in blood pressure and heart rate, nausea and vomiting, decreased blood oxygen saturation, and jaw lift) were recorded. After surgery, patients were transferred to the post-anesthesia care unit (PACU) and were allowed to return to the ward once their modified Aldrete Score reached 9.
  Interventions: Procedure: NCgroup
- SJOV group (Experimental): Received the medication regimen: propofol at 1.5-3.0 mg/kg for sedation and fentanyl at 1.5mcg/kg for analgesia. During the maintenance phase, propofol was administered via infusion at a dose of 5 mg/kg/h . The level of sedation was maintained at 0 ≤ MOAA/S score ≤ 1. When the MOAA/S score of the subjects reached 0 after induction, SJOV was administered according to the group assignment. Intraoperative vital signs were closely monitored, and data on surgery duration, anesthetic dosage, blood oxygen saturation, recovery time, and possible adverse events (significant increases or decreases in blood pressure and heart rate, nausea and vomiting, decreased blood oxygen saturation, and jaw lift) were recorded. After surgery, patients were transferred to the post-anesthesia care unit (PACU) and were allowed to return to the ward once their modified Aldrete Score reached 9.
  Interventions: Procedure: SJOVgroup

INTERVENTIONS:
Procedure: NCgroup — The patients in this group received oxygen therapy via nasal cannula at a flow rate of 5 L/min, with an oxygen concentration of 100%. An end-tidal carbon dioxide (ETCO2) monitoring catheter was placed at the nostril opening to monitor ETCO2, observe whether the waveform was regular, and record the values.
  Arms: NC group
Procedure: SJOVgroup — Gently insert an appropriately sized WNJ tube into one nostril of the subject. Connect one port of the tube to a jet ventilator (Twinstream), with the following SJOV (Synchronized Jet Ventilation) parameters: Driving pressure (DP): 15 psi (1 bar ≈ 15 psi) Respiratory rate: 15 breaths per minute Inspiratory-to-expiratory ratio (I:E): 1:2 Fraction of inspired oxygen (FiO₂): 100% Connect the other port to an end-tidal carbon dioxide (ETCO₂) monitoring catheter to observe the ETCO₂ waveform for regularity and record the numerical values.
  Arms: SJOV group

SUMMARY:
Hysteroscopic surgery is widely used in the diagnosis and treatment of gynecological diseases. Because its operation process can cause anxiety and pain in patients, it needs to be performed under anesthesia. At present, patients under conventional non-intubation general anesthesia are prone to respiratory depression and hypoxemia. Supraglottic jet oxygen supply and ventilation (SJOV) technology can provide reliable oxygen supply and ventilation for patients with respiratory arrest and respiratory depression. It can assist in completing difficult tracheal intubation, especially in emergency airway situations where "intubation and ventilation cannot be performed". It can effectively avoid catastrophic outcomes and also prevent and reduce hypoxemia in patients undergoing day surgery. However, there are very few studies on hysteroscopic surgery. This study intends to design a single-center randomized controlled study. Patients scheduled for elective hysteroscopic surgery were randomly divided into two groups: the conventional nasal catheter ventilation group and the SJOV group. The feasibility of supraglottic jet oxygenation ventilation in hysteroscopic surgery was studied through different airway management methods. The primary outcome measure was the incidence of intraoperative hypoxemia (75%≤SpO2<90%, ≤60 seconds), and the secondary outcome measures were subclinical respiratory depression, sore throat and other adverse events. The expected result is that supragttic jet ventilation can improve the incidence of hypoxia in patients during hysteroscopy, reduce sore throat or other complications at the same time, promote patient recovery, and improve patient satisfaction.

ELIGIBILITY:
inclusion criteria: Age between 18 and 65 years, with American Society of Anesthesiologists (ASA) I-II； Body mass index (BMI) between 18 and 28 kg/m²； Scheduled for elective hysteroscopic surgery under anesthesia Signed written informed consent exclusion criteria: Any upper airway abnormalities that may cause difficult airway management, such as limited mouth opening, Mallampati Class ≥ III, and abnormal neck mobility; history of respiratory insufficiency or sleep apnea, with STOP-BANG score >3; Chronic alcohol abuse or drug abuse ; Current use of anticoagulant medications; Nasal, oropharyngeal infections or other contraindications for nasopharyngeal airway/WNJ insertion, including active rhinitis, recent nasal surgery, epistaxis, nasal polyps, or nasal stenosis; Allergy to study medications ; Intraoperative conversion to endotracheal intubation due to expanded surgical scope or participant's withdrawal of consent.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxemia | Perioperative
  75%<=SPO2<90%

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Shenzhen Hospital, Guangdong, shenzhen, China

IPD SHARING:
Plan to Share IPD: No